CLINICAL TRIAL: NCT06294626
Title: Examination of Neuromotor Development of Cases Diagnosed with Scaphocephaly
Status: Completed | Type: Observational
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Ilayda Sozeri, Pediatric Physiotherapist, Acıbadem Atunizade Hospital
Other Study IDs: ISozeri
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Craniosynostosis, Sagittal; Scaphocephaly; Developmental Delay
Keywords: scaphocephaly; neuromotor development; alberta infant motor scale; denver II developmental screening test; pediatric rehabilitation
MeSH Terms: conditions — Craniosynostoses; Learning Disabilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Examination of neuromotor development of cases diagnosed with scaphocephaly: 21 cases with scaphocephaly were included. Neuromotor development was evaluated with the Denver-II Developmental Screening Test and Alberta Infant Motor Scale.
  Interventions: Other: Group 1

INTERVENTIONS:
Other: Group 1 — 21 cases with scaphocephaly diagnoses were included. Neuromotor development was evaluated with the Denver-II Developmental Screening Test and Alberta Infant Motor Scale.

SUMMARY:
It's an observational study. Purpose of the study: To evaluate the neuromotor development of scaphocephaly cases.

21 infants diagnosed with scaphocephaly aged 2-17 months were included.

* Is there any delay in the neuromotor development of scaphocephaly cases?
* If delay is observed, in which area is it most common?

Denver-II Developmental Screening Test and Alberta Motor Infant Scale were applied to the participants.

DETAILED DESCRIPTION:
Scaphocephaly (sagittal synostosis) is the most common single-suture craniosynostosis. It occurs as a result of premature ossification of the fibrous connective tissue extending between two parietal bones (sagittal suture). Phenotypically, a long and narrow head shape occurs. It occurs in 2-3 per 10,000 live births and is more common in men.

Premature ossification of the sagittal suture can lead to cranial deformity, potentially cranial growth restriction, and resulting increased intracranial pressure. In these cases, increased intracranial pressure and compression of the sagittal sinus cause increased venous pressure, which may cause developmental delays. These delays most commonly include cognitive impairments, language disorders, motor delays, learning disabilities, executive dysfunction, and behavioral problems.

When looking at the literature, it was seen that the studies were mostly on neurocognitive development in cases with craniosynostosis. There are relatively fewer studies focusing on the neuromotor development of these cases.

This study aims to evaluate the neuromotor development of scaphocephaly cases.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with scaphocephaly
* Being between 0-18 months

Exclusion Criteria:

* Be over 18 months
* Having a diagnosed disease other than scaphocephaly

Ages: 2 Months to 17 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 21 cases diagnosed with scaphocephaly aged 2-17 monts were included.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Denver-II Developmental Screening Test | baseline
  It's a screening test used in children aged 0-6 years. The test is done in a short time like 5-20 min. The person who will administer the Denver-II test; must be trained and certified. Standardized test materials are used. The test consists of 4 sections and 134 items. There are personal-social, language, fine motor and gross motor sections. The test result is classified as Normal-Abnormal-Suspicious.
Alberta Infant Motor Scale | baseline
  It's used to observe gross motor functions and evaluate the effectiveness of the intervention in typically developing infants between 0-18 months. The duration of the test is 10 min and consists of 58 items. The child's spontaneous movements are evaluated in 4 different positions without touching the child. 1 point is taken for each item that can be done. A table containing the mean and standard deviation for each month is used. The test result is classified as Normal-Abnormal-Suspicious.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.